CLINICAL TRIAL: NCT03065582
Title: The Effect of Topical Sunscreen Plus Antioxidant Against the Visible Light Biological Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Principal Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB # 9695
Record Dates: First submitted 2017-01-30; First posted 2017-02-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Pigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunscreen application (Experimental): All subjects will undergo topical application of 3 products and an additional site will serve as a control
  Interventions: Other: Topical Product A; Other: Topical Product B; Other: Topical Product C; Other: Control

INTERVENTIONS:
Other: Topical Product A — topical application sunscreen containing topical antioxidants and sunscreen filters
Other: Topical Product B — topical application of product A without topical antioxidants
Other: Topical Product C — Topical application of antioxidants only
Other: Control — No product applied

SUMMARY:
Visible light is known to induce pigmentation in darker skin types. The investigators aim to study the effects of visible light on the skin after topical application of sunscreen plus antioxidant.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 and older
* Patients Fitzpatrick skin phototype IV-VI
* Patient able to understand requirements of the study and risks involved
* Patient able to sign a consent form

Exclusion Criteria:

* A recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post inflammatory hyperpigmentation
* A known history of photodermatoses
* A known history of melanoma or non-melanoma skin cancers
* Those planning on going to the tanning parlors
* Using any of the photosensitizing medication within the visible light range or additional medications at the discretion of the investigator (examples include (but not limited to) thiazide diuretics, regular use of NSAIDs, hydroxychloroquine, or voriconazole)
* A woman who is lactating, pregnant, or planning to become pregnant
* Patient planning on exposing the irradiated or control areas to the sun
* known allergy to anesthetics (lidocaine or epinephrine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
diffuse reflectance spectroscopy | Baseline- immediately after irradiation to assess immediate pigment darkening
  Diffuse reflectance spectroscopy is a non-invasive objective measure of pigmentation based on reflectance patterns of the irradiated skin
photography | Baseline-immediately after irradiation to assess immediate pigment darkening
  Cross polarized photography is used to document pigmentation non-invasively and reduce surface glare of the skin.
investigator's global assessment score | Baseline- Immediately after irradiation to assess immediate pigment darkening
  The investigator's global assessment score is a non-invasive subjective measure of pigmentation in which investigators assign a value ranging between 0, corresponding with no hyperpigmentation, to 5, or severe or dark hyperpigmentation.
Diffuse reflectance spectroscopy | 24 hours after irradiation to assess persistent pigment darkening
  Diffuse reflectance spectroscopy is a non-invasive objective measure of pigmentation based on reflectance patterns of the irradiated skin
photography | 24 hours after irradiation to assess persistent pigment darkening
  Cross polarized photography is used to document pigmentation non-invasively and reduce surface glare of the skin.
Investigator's global assessment score | 24 hours after irradiation to assess persistent pigment darkening
  The investigator's global assessment score is a non-invasive subjective measure of pigmentation in which investigators assign a value ranging between 0, corresponding with no hyperpigmentation, to 5, or severe or dark hyperpigmentation.
Diffuse reflectance spectroscopy | 7 days after irradiation to assess delayed tanning
  Diffuse reflectance spectroscopy is a non-invasive objective measure of pigmentation based on reflectance patterns of the irradiated skin
Photography | 7 days after irradiation to assess delayed tanning
  Cross polarized photography is used to document pigmentation non-invasively and reduce surface glare of the skin.
Investigator global assessment score | 7 days after irradiation to assess delayed tanning
  The investigator's global assessment score is a non-invasive subjective measure of pigmentation in which investigators assign a value ranging between 0, corresponding with no hyperpigmentation, to 5, or severe or dark hyperpigmentation.
Biological effects | 24 hours after irradiation
  biopsy with melanocyte and melanin stains to assess pigmentation

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers.

REFERENCES:
- [Background] Mahmoud BH, Hexsel CL, Hamzavi IH, Lim HW. Effects of visible light on the skin. Photochem Photobiol. 2008 Mar-Apr;84(2):450-62. doi: 10.1111/j.1751-1097.2007.00286.x. Epub 2008 Jan 29. PMID 18248499
- [Background] Kollias N, Baqer A. An experimental study of the changes in pigmentation in human skin in vivo with visible and near infrared light. Photochem Photobiol. 1984 May;39(5):651-9. doi: 10.1111/j.1751-1097.1984.tb03905.x. No abstract available. PMID 6739557
- [Background] Porges SB, Kaidbey KH, Grove GL. Quantification of visible light-induced melanogenesis in human skin. Photodermatol. 1988 Oct;5(5):197-200. PMID 3222167
- [Background] Mahmoud BH, Ruvolo E, Hexsel CL, Liu Y, Owen MR, Kollias N, Lim HW, Hamzavi IH. Impact of long-wavelength UVA and visible light on melanocompetent skin. J Invest Dermatol. 2010 Aug;130(8):2092-7. doi: 10.1038/jid.2010.95. Epub 2010 Apr 22. PMID 20410914
- [Background] Duteil L, Cardot-Leccia N, Queille-Roussel C, Maubert Y, Harmelin Y, Boukari F, Ambrosetti D, Lacour JP, Passeron T. Differences in visible light-induced pigmentation according to wavelengths: a clinical and histological study in comparison with UVB exposure. Pigment Cell Melanoma Res. 2014 Sep;27(5):822-6. doi: 10.1111/pcmr.12273. Epub 2014 Jul 25. PMID 24888214
- [Background] Yakes FM, Van Houten B. Mitochondrial DNA damage is more extensive and persists longer than nuclear DNA damage in human cells following oxidative stress. Proc Natl Acad Sci U S A. 1997 Jan 21;94(2):514-9. doi: 10.1073/pnas.94.2.514. PMID 9012815
- [Background] Boukari F, Jourdan E, Fontas E, Montaudie H, Castela E, Lacour JP, Passeron T. Prevention of melasma relapses with sunscreen combining protection against UV and short wavelengths of visible light: a prospective randomized comparative trial. J Am Acad Dermatol. 2015 Jan;72(1):189-90.e1. doi: 10.1016/j.jaad.2014.08.023. Epub 2014 Oct 22. No abstract available. PMID 25443629
- [Background] Wang SQ, Osterwalder U, Jung K. Ex vivo evaluation of radical sun protection factor in popular sunscreens with antioxidants. J Am Acad Dermatol. 2011 Sep;65(3):525-530. doi: 10.1016/j.jaad.2010.07.009. Epub 2011 May 31. PMID 21624700
- [Background] Kunisada M, Sakumi K, Tominaga Y, Budiyanto A, Ueda M, Ichihashi M, Nakabeppu Y, Nishigori C. 8-Oxoguanine formation induced by chronic UVB exposure makes Ogg1 knockout mice susceptible to skin carcinogenesis. Cancer Res. 2005 Jul 15;65(14):6006-10. doi: 10.1158/0008-5472.CAN-05-0724. PMID 16024598
- [Background] Herrling T, Jung K, Fuchs J. Measurements of UV-generated free radicals/reactive oxygen species (ROS) in skin. Spectrochim Acta A Mol Biomol Spectrosc. 2006 Mar 13;63(4):840-5. doi: 10.1016/j.saa.2005.10.013. PMID 16543118